CLINICAL TRIAL: NCT01823679
Title: A Phase 2 Study of Capecitabine in Patients With Advanced or Recurrent Squamous Cell Carcinoma of the Skin
Brief Title: Capecitabine in Treating Patients With Advanced or Recurrent Squamous Cell Carcinoma of the Skin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A. Dimitrios Colevas, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-26699; NCI-2013-00710 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SKIN0016 (Other: OnCore)
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Squamous Cell Carcinoma of the Skin; Recurrent Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine 1000 mg/m² (Experimental): Participants will receive oral capecitabine twice-a-day (BID) as 500 mg/m² doses on days 1 to 14.
  Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda

SUMMARY:
Phase 2 evaluation of capecitabine in patients with advanced or recurrent squamous cell carcinoma of the skin.

DETAILED DESCRIPTION:
Participants are to receive 500 mg/m² of capecitabine orally (PO) twice daily (BID) on days 1 to 14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
INCLUSION CRITERIA

* Squamous cell carcinoma of the skin or "unknown primary lesions" at the time of diagnosis if metastatic disease present with a history of plausible primary skin site removed in the past. Example: squamous cell carcinoma in neck or parotid lymph nodes with no identifiable mucosal primary but with a history of the removal of one or more early stage squamous cell carcinomas of the skin in an anatomically relevant lymphatic drainage region would be eligible
* Measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension as ≥ 10 mm with computed tomography (CT) scan; magnetic resonance imaging (MRI); or calipers during clinical exam
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Life expectancy greater than 3 months
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin

  * Within normal institutional limits OR
  * ≤ 2 x upper limit of normal (ULN) if participant has Gilbert's syndrome (elevated unconjugated bilirubin from decreased UDP glucuronosyltransferase 1 family, polypeptide A1 [UGT1A1] activity)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x institutional ULN or up to 5 X ULN if known to be caused by liver metastases
* Creatinine OR

  * < 1.3 mg/dL OR
  * Creatinine clearance ≥ 30 mL/min/1.73 m2 for patients with creatinine levels above institutional normal (Note creatinine clearances between 30 and 49 mg/dL necessitate dose modification)
* For participants with a history of coronary artery disease (CAD)/myocardial infarction (MI) or congestive heart failure (CHF), ejection fraction (EF) ≥ 50% by multi-gated acquisition (MUGA) or echocardiogram (exceptions by PI discretion)

EXCLUSION CRITERIA

* Prior treatment with systemic capecitabine or prodrugs
* Prior treatment with systemic fluorouracil (5-FU) or prodrugs (prior topical treatment with 5FU is permitted if recovered from any toxicities > grade 1, and after at least 5 half-lives of the last systemically administered agent have passed)
* Receiving any other investigational agents or anti-cancer treatments
* Candidates for curative locoregional treatment (patients with recurrent locoregional disease following surgery and/ or radiation for which a resection is unacceptably morbid and unlikely to be curative are eligible)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine
* Uncontrolled concurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant
* Lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Colevas, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine 1000 mg/m²: Participants are to receive 500 mg/m² of capecitabine orally (PO) twice daily (BID) on days 1 to 14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for 2 years.
Period: Overall Study
Arm/Group | Capecitabine 1000 mg/m²
Started | 2
Completed | 1
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine 1000 mg/m²
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Response assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Time Frame: 9 weeks (3 cycles)
Measure: Number; unit: percentage of participants
Groups:
- Capecitabine 1000 mg/m²: Participants will receive oral capecitabine twice-a-day (BID) as 500 mg/m2 doses on days 1 to 14.
  Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given orally (PO)
Arm/Group | Capecitabine 1000 mg/m²
Number analyzed (Participants) | 2
percentage of participants | 0

2. Secondary Outcome: Progression-free Survival (PFS) at 1 Year
Description: Proportion of participants with progression-free survival (PFS) at 1 year, as calculated based on Kaplan-Meier estimates.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Groups:
- Capecitabine 1000 mg/m2: Participants will receive oral capecitabine twice-a-day (BID) as 500 mg/m2 doses on days 1 to 14.
  Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given orally (PO)
Arm/Group | Capecitabine 1000 mg/m2
Number analyzed (Participants) | 2
percentage of participants | 50

3. Secondary Outcome: Progression-free Survival (PFS) at 2 Years
Description: Proportion of participants with progression-free survival (PFS) at 2 years, as calculated based on Kaplan-Meier estimates.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine 1000 mg/m2
Number analyzed (Participants) | 2
percentage of participants | 0

4. Secondary Outcome: Overall Survival (OS) at 1 Year
Description: Proportion of participants with overall survival (OS) at 1 year, as calculated based on Kaplan-Meier estimates.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine 1000 mg/m2
Number analyzed (Participants) | 2
percentage of participants | 50

5. Secondary Outcome: Overall Survival (OS) at 2 Years
Description: Proportion of participants with overall survival (OS) at 2 years, as calculated based on Kaplan-Meier estimates.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine 1000 mg/m2
Number analyzed (Participants) | 2
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Capecitabine 1000 mg/m²
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine 1000 mg/m² (N=2)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Progressive Disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine 1000 mg/m² (N=2)
Hand Cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Heart Burn (Cardiac disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hand and Foot Syndrome (Infections and infestations) | 1 (1)
Nausea (General disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Weight Loss (General disorders) | 1 (1)
AST increase (Renal and urinary disorders) | 1 (1)
Alk P'Tase increase (Renal and urinary disorders) | 1 (1)
Dysguesia (Gastrointestinal disorders) | 1 (1)
Rash (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No